CLINICAL TRIAL: NCT01284426
Title: The Natural History of Chronic Urticaria in Childhood: A Prospective Study
Brief Title: Natural History of Chronic Urticaria
Acronym: NHCU
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Prof., Mahidol University
Other Study IDs: 374/2551(EC3)
Record Dates: First submitted 2011-01-20; First posted 2011-01-27 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria; Natural course; Remission
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic urticaria: Chronic urticaria, Natural history

SUMMARY:
The purpose of this study is to examine the natural history of chronic urticaria in children and to identify the predictors for chronic urticaria remission.

DETAILED DESCRIPTION:
A Prospective cohort study of 92 children who were diagnosed with chronic urticaria to investigate the natural course of chronic urticaria and to identify predictors of disease remission.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-15 years of age with the diagnosis of chronic urticaria who were attending the pediatric allergy clinic, Siriraj Hospital Mahidol University, Thailand, from March 2003 to March 2009.

Exclusion Criteria:

* Children who had isolated physical urticaria, inability to be followed up, pregnancy, underlying diseases such as cardiovascular, hepatobiliary, and renal diseases.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric allergy clinic, Siriraj Hospital Mahidol University, Thailand, Children 4-15 years of age with chronic urticaria.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2003-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, Prof., Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Chansakulporn S, Pongpreuksa S, Sangacharoenkit P, Pacharn P, Visitsunthorn N, Vichyanond P, Jirapongsananuruk O. The natural history of chronic urticaria in childhood: a prospective study. J Am Acad Dermatol. 2014 Oct;71(4):663-8. doi: 10.1016/j.jaad.2014.05.069. Epub 2014 Jul 11. PMID 25023899
- See also: The natural history of chronic urticaria in childhood: a prospective study. — http://www.ncbi.nlm.nih.gov/pubmed/?term=J+Am+Acad+Dermatol.+2014+Oct%3B71(4)%3A663-8.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Urticaria
Started | 94
Completed | 92
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Remission period, chronic urticaria
Arm/Group | Chronic Urticaria
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: Years] — Children 4-15 years of age
  Years | 8.4 [4.0 to 15.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 43
Region of Enrollment [Number; unit: participants]
  Thailand | 92

OUTCOME MEASURES:

1. Primary Outcome: Duration of Urticaria Until Remission Since Chronic Urticaria Was Diagnosed.
Description: Remission rates at 1, 3 and 5 years after the onset of symptoms of chronic urticaria.
  Description in details:
  Actually, this study have been started in March 2003 and finally done in March 2009, which would be totally 6 years. We eventually decided to report the rate of CU remissions only at 1, 3 and 5 years after the onset of symptoms because this would be the common interval time of CU symptoms that patients needed to know how long they should have those CU symptoms or how many of them would go away their symptoms within 1, 3 or 5 years. Another reason is that the remission rate of CU between 5 and 6 years was not significantly different, so it might not need to be reported.
Time Frame: 6 years
Population: Children 4-15 years old with chronic urticaria
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Urticaria
Number analyzed (Participants) | 92
percentage of participants
  Remission rate at 1 year after the onset | 18.5
  Remission rate at 3 year after the onset | 54
  Remission rate at 5 year after the onset | 67.7

ADVERSE EVENTS:
Time Frame: 6 years. Actually, this study is the prospective observational study of chronic urticaria for over 6 years regarding only the remission of the disease.
Description: Since we did not add any intervention into the participants, therefore, we did not observe any serious or non-serious adverse events other than the activity or remission of chronic urticaria. However, if we consider as the Total Number of Participants at Risk, the number should be "92 participants" or "100%".
Arm/Group | Chronic Urticaria
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 62/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Urticaria (N=92)
Remission of chronic urticaria after 1 year of symptoms (Skin and subcutaneous tissue disorders) | 17 (17) — Remission of chronic urticaria (CU) after 1 year of the onset of symptoms was considered if symptoms did not recur for at least 12 months without medication after 1 years of CU symptoms.
Remission of chronic urticaria after 3 years of symptoms (Skin and subcutaneous tissue disorders) | 50 (50) — Remission of chronic urticaria (CU) after 3 years of the onset of symptoms was considered if symptoms did not recur for at least 12 months without medication after 3 years of CU symptoms.
Remission of chronic urticaria (CU) after 5 years of symptoms (Skin and subcutaneous tissue disorders) | 62 (62) — Remission of chronic urticaria (CU) after 5 years of the onset of symptoms was considered if symptoms did not recur for at least 12 months without medication after 5 years of CU symptoms.

LIMITATIONS AND CAVEATS:
This study did not perform basophil histamine releasing assay to identify the existence of functional autoantibodies, since there was no available laboratory to do this test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No